CLINICAL TRIAL: NCT00120848
Title: Study of the Efficacy of Candidate HPV 16/18 VLP Vaccine in the Prevention of HPV-16 and/or HPV-18 Cervical Infection in Adolescent & Young Adult Women in North America and Brazil Vaccinated in Primary Study 580299/001
Brief Title: Follow-up Study of GSK Biologicals' Human Papilloma Virus (HPV) Vaccine to Prevent Cervical Infection in Young Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 580299/007
Record Dates: First submitted 2005-07-12; First posted 2005-07-19 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Infections, Papillomavirus
Keywords: HPV vaccine efficacy; Prophylaxis HPV 16/18 infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Biological: HPV 16/18 VLP AS04

SUMMARY:
Human Papilloma virus (HPV) are viruses that cause a common infection of the skin and genitals in men and women. Several types of HPV infection are transmitted by sexual activity and, in women, can infect the cervix (part of the uterus or womb). This infection often goes away by itself, but if it does not go away (this is called persistent infection), it can lead in women over a long period of time to cancer of the cervix. If a woman is not infected by HPV, it is very unlikely that she will get cervical cancer. This is an observer blind follow up study of the study HPV-001, which evaluated the ability of the HPV vaccine to prevent HPV infection. The current study invites all of the 1113 subjects in the HPV-001 study that received all three doses of vaccine/placebo to be enrolled and followed-up for several additional years to see if the HPV vaccine prevents HPV-16 and HPV-18 infections and to evaluate the safety of the vaccine. Subjects will remain in the same study group as in the primary study. No vaccine or placebo will be administered in this study.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Participated in study 580299/001 and received all three doses of vaccine/placebo.
* Written informed consent obtained from the subject prior to enrollment

Exclusion Criteria:

* Decoding of the subject's treatment allocation to either the subject or the investigator in study 580299/001.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 776 (Actual)
Dates: Start 2003-11; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Incident cervical infection with HPV-16 and/or HPV-18

SECONDARY OUTCOMES:
Persistent cervical infection (6-month definition) with HPV 16 and/or HPV 18.
Persistent cervical infection (6-month definition) with oncogenic HPV types.
Incident cervical infection with oncogenic HPV types.
Histopathologically-confirmed CIN 1+ or CIN 2+ associated with HPV 16 and/or HPV 18 detected within the lesional component of the cervical tissue specimen.
Histopathologically-confirmed CIN 1+ or CIN 2+ associated with oncogenic HPV types detected within the lesional component of the cervical tissue specimen.
Abnormal cytology associated with an HPV-16 and/or HPV-18 cervical infection.
Abnormal cytology associated with oncogenic HPV type cervical infection.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- United States (16):
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, Lebanon, New Hampshire
  - GSK Investigational Site, Morristown, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Marshfield, Wisconsin
- Brazil (5):
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, São Paulo, São Paulo
  - GSK Investigational Site, Campinas
  - GSK Investigational Site, Fortaleza
- Canada (5):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Langley, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, St. John's, Newfoundland and Labrador
  - GSK Investigational Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] David MP, Van Herck K, Hardt K, Tibaldi F, Dubin G, Descamps D, Van Damme P. Long-term persistence of anti-HPV-16 and -18 antibodies induced by vaccination with the AS04-adjuvanted cervical cancer vaccine: modeling of sustained antibody responses. Gynecol Oncol. 2009 Dec;115(3 Suppl):S1-6. doi: 10.1016/j.ygyno.2009.01.011. Epub 2009 Feb 12. PMID 19217149
- [Background] Descamps D, Hardt K, Spiessens B, Izurieta P, Verstraeten T, Breuer T, Dubin G. Safety of human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine for cervical cancer prevention: a pooled analysis of 11 clinical trials. Hum Vaccin. 2009 May;5(5):332-40. doi: 10.4161/hv.5.5.7211. Epub 2009 May 20. PMID 19221517
- [Background] Harper DM, Franco EL, Wheeler CM, Moscicki AB, Romanowski B, Roteli-Martins CM, Jenkins D, Schuind A, Costa Clemens SA, Dubin G; HPV Vaccine Study group. Sustained efficacy up to 4.5 years of a bivalent L1 virus-like particle vaccine against human papillomavirus types 16 and 18: follow-up from a randomised control trial. Lancet. 2006 Apr 15;367(9518):1247-55. doi: 10.1016/S0140-6736(06)68439-0. PMID 16631880
- [Background] Katherine A et al. (2012) Adjuvanted human papillomavirus types 16/18 vaccine (Cervarix®): a guide to its use. Adis Drug Eval Drug Prof. 28(3):1-6.
- [Background] GlaxoSmithKline Vaccine HPV-007 Study Group; Romanowski B, de Borba PC, Naud PS, Roteli-Martins CM, De Carvalho NS, Teixeira JC, Aoki F, Ramjattan B, Shier RM, Somani R, Barbier S, Blatter MM, Chambers C, Ferris D, Gall SA, Guerra FA, Harper DM, Hedrick JA, Henry DC, Korn AP, Kroll R, Moscicki AB, Rosenfeld WD, Sullivan BJ, Thoming CS, Tyring SK, Wheeler CM, Dubin G, Schuind A, Zahaf T, Greenacre M, Sgriobhadair A. Sustained efficacy and immunogenicity of the human papillomavirus (HPV)-16/18 AS04-adjuvanted vaccine: analysis of a randomised placebo-controlled trial up to 6.4 years. Lancet. 2009 Dec 12;374(9706):1975-85. doi: 10.1016/S0140-6736(09)61567-1. PMID 19962185
- [Background] Schwarz TF et al. (2011) Overview of clinical evidence: Cervarix. Future Medicine - Human Papillomavirus Vaccines. 38-50.
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- [Derived] El-Zein M, Ramanakumar AV, Naud P, Roteli-Martins CM, de Carvalho NS, Colares de Borba P, Teixeira JC, Moscicki AB, Harper DM, Tyring SK, Ramjattan B, Dubin G, Franco EL; HPV-007 Study Group. Determinants of Acquisition and Clearance of Human Papillomavirus Infection in Previously Unexposed Young Women. Sex Transm Dis. 2019 Oct;46(10):663-669. doi: 10.1097/OLQ.0000000000001053. PMID 31464859
- [Derived] Ramanakumar AV, Naud P, Roteli-Martins CM, de Carvalho NS, de Borba PC, Teixeira JC, Blatter M, Moscicki AB, Harper DM, Romanowski B, Tyring SK, Ramjattan B, Schuind A, Dubin G, Franco EL; HPV-007 Study Group. Incidence and duration of type-specific human papillomavirus infection in high-risk HPV-naive women: results from the control arm of a phase II HPV-16/18 vaccine trial. BMJ Open. 2016 Aug 26;6(8):e011371. doi: 10.1136/bmjopen-2016-011371. PMID 27566633
- [Derived] Naud PS, Roteli-Martins CM, De Carvalho NS, Teixeira JC, de Borba PC, Sanchez N, Zahaf T, Catteau G, Geeraerts B, Descamps D. Sustained efficacy, immunogenicity, and safety of the HPV-16/18 AS04-adjuvanted vaccine: final analysis of a long-term follow-up study up to 9.4 years post-vaccination. Hum Vaccin Immunother. 2014;10(8):2147-62. doi: 10.4161/hv.29532. PMID 25424918
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 580299/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 580299/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 580299/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 580299/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 580299/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 580299/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 580299/007 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register